CLINICAL TRIAL: NCT04490486
Title: Phase I, Randomized, Double Blinded, Placebo Control Study to Evaluate the Safety and Potential Efficacy of Intravenous Infusion of Umbilical Cord Tissue (UC) Derived Mesenchymal Stem Cells (MSCs) Versus Placebo to Treat Acute Pulmonary Inflammation Due to COVID-19 With Moderate to Severe Symptoms
Brief Title: Umbilical Cord Tissue (UC) Derived Mesenchymal Stem Cells (MSCs) Versus Placebo to Treat Acute Pulmonary Inflammation Due to COVID-19
Acronym: COVID-19
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not Funded
Sponsor: Joshua M Hare (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Director of ISCI, Louis Lemberg Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20200575
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome; Corona Virus Infection
Keywords: Acute Pulmonary Inflammation
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: (UCMSCs) (Experimental): Participants in this group will receive the 2 intravenous (IV) UCMSCs intervention on day 0 and day 3.
  Interventions: Biological: UCMSCs
- Group 2: (Placebo) (Placebo Comparator): Participants in this group will receive the placebo, a solution of 1% human serum albumin in Plasmalyte A, on day 0 and day 3.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: UCMSCs — 100 x 106 (100 million) UCMSCs delivered via peripheral intravenous infusion.
  Arms: Group 1: (UCMSCs)
Other: Placebo — Placebo, a solution of 1% human serum albumin in Plasmalyte A, delivered via peripheral intravenous infusion
  Arms: Group 2: (Placebo)

SUMMARY:
The purpose of this study is to demonstrate the safety of Umbilical Cord Tissue Derived Mesenchymal Stem Cells (UCMSCs) administered intravenously in patients with acute pulmonary inflammation due to COVID-19 with moderately severe symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Male or female subjects age > 18 years at the time of signing the Informed Consent Form.
3. COVID-19 positive according to diagnosis (evaluated by reverse transcription (RT)-polymerase chain reaction (PCR) test confirming infection with severe acute respiratory syndrome coronavirus and clinical management of COVID-19 criteria (refer to appendix B)
4. Individuals with moderate to severe COVID-19 symptoms.

   * Moderate:
   * Patients with moderate disease are symptomatic (e.g. fever, cough, headache, myalgia, sore throat, nasal congestion, nausea, vomiting, diarrhea, fatigue, anosmia, or dysgeusia) and have abnormal chest imaging or some degree of hypoxia requiring supplemental oxygen but not intubation.
   * Moderate-severe:
   * The Moderately Severe disease category includes patients who are symptomatic (as described above), have abnormal chest imaging, but also have worsening hypoxia compatible with mild acute respiratory distress syndrome (ARDS) (Partial Pressure of Oxygen (PaO2)/Fraction of Inspired Oxygen (FiO2) </= 300 but > 200) - Berlin criteria; but do not yet require intubation .
5. Adequate venous access
6. For female patients only, willingness to use FDA-recommended birth control until 6 months post treatment.
7. Must agree to comply with all study requirements and be willing to complete all study visits.
8. Need in-patient admission

Exclusion Criteria:

1. PaO2/FiO2 </= 200
2. Anticipated intubation within 24h
3. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood pregnancy test at screening and prior to infusion.
4. Inability to perform any of the assessments required for endpoint analysis.
5. Subjects that are unsuitable with the study requirements .
6. Active listing (or expected future listing) for transplant of any organ.
7. Have known allergies to penicillin or streptomycin.
8. Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior to enrollment), bone, skin, ligament, tendon or corneal grafting.
9. Have a history of organ or cell transplant rejection
10. Has a history of an adverse response to cell-based therapy
11. Have presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the last 1 year.
12. History of active drug abuse (illegal "street" drugs except marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months
13. Be serum positive for HIV, Surface antigen of Hepatitis B virus (HBsAg) or Viremic hepatitis C.
14. Severe hepatic impairment (defined as liver cirrhosis Child stage B or C);
15. Stage 4 chronic kidney disease or currently receiving chronic dialysis;
16. Advanced cardiac (eg, severe heart failure [New York Heart Association (NYHA) III-IV]) or pulmonary diseases;
17. Has uncontrolled hypertension as defined by BP systolic above 180 and diastolic above 110 which, in the Investigator's judgment, would not make participation appropriate;
18. Known allergy or hypersensitivity to stem cell infusions or its components;
19. Current enrollment in an investigational drug or participation in such a study within 15 days of entry into this study;
20. Moderate to severe liver failure (Childs-Pugh Score > 10) Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) > 5 times the upper limit of normal;
21. Congenital prolonged QT syndrome;
22. Current QT corrected (QTc) above 490 msec. If patient has Q, R and S waves (QRS) interval greater or equal to 120 msec, then the QT/QTc will be normalized to a QRS interval of 110 msec. (For instance, if the patient has a bundle branch block with QRS of 140 msec and QT/QTc of 470 msec, the normalized QTc will be 470;
23. Subjects taking drugs that could affect the QT interval (e.g. procainamide, disopyramide, mexiletine, flecainide, propafenone, amiodarone, sotalol, cimetidine, dronedarone, dofetilide, levofloxacin, ciprofloxacin, moxifloxacin);
24. Anticipated transfer to another hospital which is not a study site within 72 hours;
25. Coagulopathy (Platelets less than 80,000, or Prothrombin Time (PT)/Partial Thromboplastin time (PTT) twice normal range without systemic anticoagulation;
26. Greater than 24h since first meeting ARDS criteria (Berlin definition) or 72h of ICU admission;
27. Subjects who are legally detained in an official institution;
28. A previous MSC infusion in last 30 days not related to this trial;
29. History of Pulmonary Hypertension (WHO Class III/IV);
30. Unstable arrhythmia or uncontrolled hypertension not responding to best ICU treatment;
31. Patients currently receiving Extracorporeal Membrane Oxygenation (ECMO);
32. Any other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%;
33. Moribund patient not expected to survive > 24 hours;
34. The investigator believes that participating in the trial is not in the best interest of the patient, or the investigator considers patient unsuitable for enrollment (such as unpredictable risks or subject compliance issues)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with treatment related Serious Adverse Events (SAE) | 12 months
  Safety of UCMSCs will be reported as the percentage of participants in each treatment group that experienced a treatment related SAEs.

SECONDARY OUTCOMES:
Change in inflammatory marker levels | Baseline, Day 30
  Change in serum inflammatory marker levels including Interleukin (IL) IL-6, IL-2, Tumor Necrosis Factor Alpha (TNF-a) and procalcitonin will be evaluated in ng/L.
Change in systemic inflammatory marker levels | Baseline, Day 30
  Change in serum systemic inflammatory marker levels including D-dimer, high sensitivity C-reactive protein (hsCRP) and ferritin will be evaluated in mg/L.
COVID-19 Viral Load | Up to 30 Days
  Assessed using blood samples or nose/throat swabs.
Change in SOFA score | Baseline, Up to 30 Days
  Sequential Organ Failure Assessment (SOFA) will be used to assess organ failure including the cardiovascular system, coagulation system, liver, kidney and other extra-pulmonary organs. SOFA score ranges from 0-24 with the higher score indicating worse outcomes.
Change in electrolytes levels | Baseline, Up to 30 Days
  Sodium, Potassium, Chloride and Carbon Dioxide (CO2) will be evaluated in mmol/L. Changes from baseline to Day 30 will be compared between groups.
Change in LDH levels | Baseline, Up to 30 Days
  Serum Lactate Dehydrogenase (LDH) levels assessed in U/L. Changes in LDH from baseline to Day 30 will be compared between groups.
Number of subjects discharged from the ICU | Up to 7 Days
  ICU monitoring status will be reported as the number of subjects discharged from the ICU within 7 days.
Percentage of participants with less requirement for vasoactive agents | Up to 30 Days
  Percentage of participants requiring less use of vasoactive agents will be reported.
Rate of Mortality | Up to 30 Days
  Percentage of participant deaths throughout the study period.
Percentage of participants with changes in immune marker expression | Up to 30 Days
  The percentage of participants with changes in serum immune marker levels including Cluster of Differentiation (CD) CD 4+ and CD 8+, as evaluated by treating physician will be reported.
Percentage of participants with changes in radiologic findings | Up to 30 Days
  Percentage of participants with changes in their chest imaging such as ground-glass opacity, local patch shadowing, bilateral patch shadowing and interstitial abnormalities will be reported. Imaging will be assessed by treating physician using chest radiography or chest Computed Tomography (CT).
Percentage of participants with less pneumonia symptoms | Up to 30 Days
  Percentage of participants showing less pneumonia symptoms will be reported as evaluated by treating physician using chest radiography or chest CT.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — ISCI/University of Miami Miller School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interdisciplinary Stem Cell Institute at the University of Miami Miller School website — http://isci.med.miami.edu/